CLINICAL TRIAL: NCT07193017
Title: The Effects of Biphasic Positive Airway Pressure (BIPAP) Use on Diaphragm Functions in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: The Effect of BIPAP on Diaphragmatic Function
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Demiroglu Bilim University (Other)
Collaborators: Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Reyhan Kaygusuz, Assistant Professor, Istanbul Demiroglu Bilim University
Other Study IDs: Effect of BIPAP on diaphragm
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: BIPAP Biphasic Intermittent Positive Airway Pressure; Diaphragm Issues; Ultrasound Diagnostics; COPD (Chronic Obstructive Pulmonary Disease)
Keywords: bıpap, diaphragm function, diaphragm ultrasound, copy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- copd patients: Patients diagnosed with chronic obstructive pulmonary disease (COPD) who have been prescribed BiPAP therapy by a physician. Participants will undergo diaphragmatic function evaluations with ultrasound at baseline, after 6 weeks of BiPAP usage, and after one year.
  Interventions: Device: BIPAP

INTERVENTIONS:
Device: BIPAP — After BIPAP Prescribed By A Physician, Diaphragmatic Functions Will Be Evaluated With Ultrasound In The Early And Late Periods

SUMMARY:
This research is designed to evaluate how long-term treatment with Bilevel Positive Airway Pressure (BiPAP) influences diaphragm function in patients with Chronic Obstructive Pulmonary Disease (COPD) who suffer from chronic hypercapnic respiratory failure. The diaphragm is the primary muscle of breathing, and its dysfunction is linked to unfavorable clinical outcomes such as higher mortality rates and frequent hospitalizations. In this prospective cohort study, COPD patients starting BiPAP therapy based on clinical indication will be monitored through repeated ultrasound assessments of diaphragm structure and function together with pulmonary function testing, respiratory muscle strength evaluation, dyspnea. The main outcome of interest is the change in diaphragm thickness in inspiration, thickness in expiration, diaphragm thickening fraction (DTF), diaphragm maximum contraction velocity and maximum relaxation velocity across a 6 weeks as a early time and 12 months for long time follow-up period. Secondary measures include hospital admissions, and one-year survival. The study is expected to generate valuable evidence about the link between non-invasive ventilation and diaphragm function, which may contribute to optimizing treatment strategies for COPD patients with advanced respiratory failure.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a progressive respiratory condition frequently complicated by chronic hypercapnic respiratory failure. In this population, long-term non-invasive ventilation with bilevel positive airway pressure (BiPAP) is widely prescribed to improve gas exchange, relieve symptoms, and reduce the risk of hospitalizations. However, its effects on diaphragm function, the main respiratory muscle, remain poorly understood. Diaphragm dysfunction in COPD has been associated with adverse outcomes including increased mortality, prolonged hospital stay, and higher readmission rates.

This prospective cohort study aims to evaluate the longitudinal impact of BiPAP treatment on diaphragm structure and function in patients with COPD and chronic hypercapnic respiratory failure. Eligible participants will be patients who are prescribed BiPAP therapy according to standard clinical indications. Diaphragm function will be assessed repeatedly using ultrasonography, which provides non-invasive and reliable measurements of diaphragm thickness at end-inspiration and end-expiration, thickening fraction (DTF), maximum contraction velocity, and maximum relaxation velocity. These measurements will be complemented by pulmonary function tests, respiratory muscle strength evaluations, and dyspnea assessment.

The primary outcome is the change in diaphragm ultrasound parameters (inspiratory thickness, expiratory thickness, thickening fraction, contraction velocity, and relaxation velocity) over the course of treatment. Early follow-up will occur at 6 weeks to assess short-term effects, while long-term follow-up at 12 months will provide insight into sustained adaptations to BiPAP therapy. Secondary outcomes include the frequency of hospital admissions and overall one-year survival.

By integrating functional, structural, and clinical outcomes, the study is expected to provide novel evidence on the role of non-invasive ventilation in modifying diaphragm performance. Findings may contribute to refining treatment strategies and optimizing long-term management of COPD patients with advanced respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Being between 40-80 years of age,
* Having a diagnosis of stable COPD for at least 1 year,
* Being in a stable phase (no acute exacerbation within the last 4 weeks),
* Meeting the GOLD 2025 A-B-E classification according to symptoms and exacerbation history,
* Having been initiated on BiPAP therapy with a clinical indication,
* Being willing to participate in the study and providing informed consent.

Exclusion Criteria:

* Pregnancy,
* Diaphragmatic paralysis,
* Neuromuscular and neurological diseases,
* Decompensated heart failure,
* Chest deformity,
* Acute exacerbation within the last month,
* Pneumothorax,
* Body mass index greater than 35 kg/m²,
* Long-term corticosteroid use,
* Chemotherapy,
* Active malignancy,
* Inability to cooperate,
* Thoracoabdominal surgery within the last 3 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patient prescribed BIPAP
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
One-Year Survival | at baseline and after 12 months
  Survival status (alive or deceased) will be assessed at 12 months after initiation of BiPAP therapy. This will be recorded as a binary outcome.
Number of Hospital Admissions within 12 Months | at baseline and after 12 months
  The number of hospital admissions due to respiratory or other causes will be recorded during the 12-month follow-up period. A higher number indicates greater healthcare utilization.
Maximum Inspiratory Pressure (MIP) | Baseline, after 6 weeks of BiPAP usage, and after one year
  Respiratory muscle strength will be assessed using maximum inspiratory pressure (MIP), measured with a portable mouth pressure device according to standard guidelines. Higher values indicate better inspiratory muscle function.
Maximum Expiratory Pressure (MEP) | At baseline, after 6 weeks of BiPAP usage, and after one year.
  Respiratory muscle strength will be assessed using maximum expiratory pressure (MEP), measured with a portable mouth pressure device according to standard guidelines. Higher values indicate better expiratory muscle function.
Forced Vital Capacity (FVC) | Baseline, after 6 weeks of BiPAP usage, and after one year.
  Forced Vital Capacity (FVC) will be measured using a portable spirometer calibrated according to American Thoracic Society (ATS) and European Respiratory Society (ERS) standards. The best result from at least three attempts will be recorded.
Forced Expiratory Volume in 1 Second (FEV₁) | Baseline, after 6 weeks of BiPAP usage, and after one year.
  Forced Expiratory Volume in 1 second (FEV₁) will be measured using a portable spirometer calibrated according to ATS/ERS standards. The best result from at least three attempts will be recorded.
FEV₁/FVC Ratio | Baseline, after 6 weeks of BiPAP usage, and after one year.
  FEV₁/FVC ratio will be calculated from spirometry results. The best result from at least three attempts will be recorded.
Cough Strength (Peak Cough Flow, PCF) | Baseline, after 6 weeks of BiPAP usage, and after one year.
  Peak Cough Flow (PCF) will be measured using a peak flow meter.
Diaphragm Thickness (B-mode Ultrasound) | Baseline, after 6 weeks of BiPAP usage, and after one year.
  Diaphragm thickness will be measured in two-dimensional B-mode ultrasound from the right intercostal area (mid-axillary level), the right subcostal area (anterior axillary level and mid-clavicular level) with a superficial probe during deep inspiration and deep expiration.
Diaphragm Excursion (M-mode Ultrasound) | Baseline, after 6 weeks of BiPAP usage, and after one year.
  Diaphragm mobility during normal inspiration and deep inspiration will be assessed using M-mode ultrasonography from the right subcostal area at the mid-axillary level.
Diaphragmatic Tissue Velocity (Tissue Doppler Imaging) | Baseline, after 6 weeks of BiPAP usage, and after one year.
  Diaphragmatic tissue waveform and movement velocities during inspiration and expiration will be assessed using tissue Doppler ultrasonography. Maximum contraction and relaxation rates of the diaphragm will be recorded during 10 normal breaths.

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) Score: | at baseline and after 6 weeks of BIPAP usage and after one year
  CAT will be used to assess health status impairment in patients with respiratory symptoms. Higher scores indicate greater symptom burden.
Dyspnea (mMRC Scale) | at baseline and after 6 weeks of BIPAP usage and after one year
  Dyspnea severity will be evaluated using the modified Medical Research Council (mMRC) dyspnea scale, ranging from 0 (no dyspnea) to 4 (severe dyspnea).

CONTACTS AND LOCATIONS:
Overall Officials: Reyhan Kaygusuz Benli, Asst Prof, Principal Investigator — Demiroglu Bilim University, Dept. of Physiotherapy and Rehabilitation
Locations (1):
- Demiroglu Bilim University, Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No